CLINICAL TRIAL: NCT02958163
Title: Randomized Controlled Phase II Trial Comparing Trans-Arterial Chemo-Embolization (TACE) With TACE Plus Stereotactic Ablative Radiotherapy (SABR) in Stage BCLC B Hepatocarcinoma (HepSTAR)
Brief Title: Clinical Trial Comparing TACE With TACE + SABR in Stage BCLC B HCC (HepSTAR)
Acronym: HepSTAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Erasme University Hospital (Other); Jules Bordet Institute (Other); University of Liege (Other); Clinique Saint Joseph, Liège (Other); Centre Hospitalier Universitaire UCLouvain Namur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28248368
Record Dates: First submitted 2016-10-26; First posted 2016-11-08 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-03

CONDITIONS: Liver Neoplasms; Hepatocellular Cancer
Keywords: Hepatocellular cancer; Stereotactic Body Radiotherapy; Chemoembolization, Therapeutic
MeSH Terms: conditions — Liver Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-Arterial Chemo-embolization (TACE) (Active Comparator): Trans-arterial Embolisation will be performed with drug-eluting beads loaded with Doxorubicin. First session will be given within 4 weeks after randomization.
  4-phase MRI will be performed every 2 months to assess the response. In case of insufficient response according to the MRI performed at 2 or 4 months, a second or third session of DEB-TACE will be allowed, according to the physician's choice.
  Once complete response is achieved, the follow-up period will start. The date of the last session of TACE corresponds to the treatment completion date.
  Interventions: Procedure: Trans-arterial Chemo-Embolization; Drug: Doxorubicin
- TACE+Stereotactic Ablative Radiotherapy (Experimental): The first part of the treatment, which is the DEB-TACE delivery, will be exactly the same than in arm A. The radiotherapy (SABR) will then start within 4 to 6 weeks after.
  Afterwards, 4-phase MRI will be performed every 2 months to assess the response. In case of insufficient response according to the MRI performed at 2 or 4 months, a second or third session of DEB-TACE will be allowed, according to the physician's choice.
  Once complete response is achieved, the follow-up period will start. The date of the last SABR fraction or the last session of TACE corresponds to the treatment completion date.
  Interventions: Procedure: Trans-arterial Chemo-Embolization; Drug: Doxorubicin; Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Procedure: Trans-arterial Chemo-Embolization — Trans-Arterial Chemo-Embolization will be performed with Doxorubicin-Eluting-Beads (DEB-TACE). It will be performed in each arm of treatment.
  Other Names: TACE
Drug: Doxorubicin — Drug-eluting Bead for Trans Arterial Chemo-Embolization will be loaded with Doxorubicin.
  Other Names: DEB-TACE
Radiation: Stereotactic Ablative Radiotherapy — SABR schemes will be adapted according to the CP score and the vicinity of surrounding organs at risk. These are the different schemes proposed in this trial:
  48Gy = 3x16Gy BED 124.8Gy ( α/β=10) 50Gy = 5x10Gy BED 100Gy ( α/β=10) 48Gy = 6x8Gy BED 86.4Gy ( α/β=10) 40Gy = 5x8Gy BED 72Gy ( α/β=10)
  For patients with Child-Pugh (CP) A cirrhosis : the choice of the scheme will be left to each physician. The highest BED should be favored if dose constraints to the organs at risk are respected.
  For patients with CP B cirrhosis : only the latter scheme will be allowed: 40Gy = 5x8Gy.
  Other Names: SABR
  Arms: TACE+Stereotactic Ablative Radiotherapy

SUMMARY:
This will be multicentre a phase II randomized controlled and open-label trial. It will compare the 6-months objective response (CR+PR) rates obtained with Drug Eluting Bead Trans-Arterial Chemo-Embolization (DEB-TACE) alone versus DEB-TACE followed by Stereotactic Ablative Radiotherapy (SABR) in patients with hepatocarcinoma stage BCLC B.

This trial will also include one substudy. This substudy will confront the immuno-histochemical results collected on tumoral biopsies to the biological and imaging (MRI) results. Every patient participating to the trial can also participate to this substudy.

DETAILED DESCRIPTION:
The patients will be randomized in 2 arms determining the treatment they will receive:

Arm A: actual standard treatment = TACE Arm B: experimental arm = TACE + SABR

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma larger than 3 cm and non-resectable, with a diagnosis established either by:

  * dynamic imaging (non-invasively), showing a typical contrast enhancement and wash-out
  * histopathology
* satellite lesions are allowed (at most three lesions) as long as the doses constraints are still achievable
* Hepatocellular carcinoma belonging to Barcelona Clinic Liver Cancer Stage System class B
* Tumor must be measurable on a multi-phase MRI according to mRECIST criteria
* Non-tumoral liver volume ≥ 800 cc
* Child-Pugh (CP) A to B7 cirrhosis
* HCC Patients can be included if they require treatment prior to liver transplantation
* ECOG performance status 0-1
* AST/ALT < 5 times ULN
* Initial platelets ≥ 50 000 x 10E9/l, neutrophils > 1500 x 10E9/l, Hb > 9 g/dl
* Serum creatinine < 1.5 X normal, or calculated Creatinine clearance rate ≥ 60 mL/min
* As tumor biopsy can be performed after inclusion, pure hepatocellular carcinoma but also mixed hepatocellular carcinoma will be allowed in this trial. Cholangiocarcinoma cannot be included.
* Written informed consent form to be signed,
* Patient willing and able to comply to the follow-up schedule
* Patients in fertile age should use a contraceptive method during treatment and 4 months after.

Exclusion Criteria:

* Eligibility for resection or ablative treatments
* Extra hepatic spread of the disease
* Previous treatment of the same lesion with TACE
* Previous treatment with selective internal radiotherapy or radiotherapy to the upper abdomen
* Uncontrolled Ascites
* Uncontrolled Encephalopathy
* Any clinical sign of acute viral or non-viral hepatitis (new serological testing are not required)
* Known current pregnancy
* Uncontrolled active co-morbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Objective response rate at 6 months | 6 months after the completion of treatment
  Objective response rate including complete and partial response based on the MRI evaluation (mRECIST)

SECONDARY OUTCOMES:
Time to progression | 1 year after the treatment completion
  defined as the time between the end of treatment and the occurrence of a local recurrence. The diagnoses of another intra- or extra-hepatic lesion of HCC will not be considered as progression
Time to untreatable progression | 1 year after the treatment completion
  defined as the time between the end of treatment and the occurrence of untreatable intra-hepatic disease
6-months overall survival | 1 year after the treatment completion
  defined as survival rate of patients at 6months after the end of treatment
1-year overall survival | 1 year after the treatment completion
  defined as survival rate of patients at 1 year after the end of treatment
Acute toxicities | 6 months after treatment completion
  Acute toxic events will have to be described and recorded in accordance with the CTCAE 4.03 (Common Terminology Criteria for Adverse events).
Late toxicities | 6 months after treatment completion
  Late toxic events will have to be described and recorded in accordance with the CTCAE 4.03 (Common Terminology Criteria for Adverse events).
Quality of life assessment by questionnaire at baseline | baseline
  Quality of life will be assessed by questionnaires: EORTC QLQC30. The investigators will ask each patient to answer to these questionnaires once at randomization.
Quality of life assessment by questionnaire at 2 months | 2 months
  Quality of life will be assessed by questionnaires: EORTC QLQC30. The investigators will ask each patient to answer to these questionnaires 2 months after treatment completion
Quality of life assessment by questionnaire at 6 months | 6 months after treatment completion
  Quality of life will be assessed by questionnaires: EORTC QLQC30. The investigators will ask each patient to answer to these questionnaires 6 months after treatment completion
Assessment by questionnaires of specific for hepatocarcinoma quality of life at baseline | baseline
  Quality of life will be assessed by questionnaires specific for patients with hepatocarcinoma:EORTC QLQH18. The investigators will ask each patient to answer to these questionnaires once at randomization.
Assessment by questionnaires of specific for hepatocarcinoma quality of life at 2 months | 2 months after treatment completion
  Quality of life will be assessed by questionnaires specific for patients with hepatocarcinoma:EORTC QLQH18. The investigators will ask each patient to answer to these questionnaires 2 months after treatment completion
Assessment by questionnaires of specific for hepatocarcinoma quality of life at 6 months | 6 months after treatment completion
  Quality of life will be assessed by questionnaires specific for patients with hepatocarcinoma:EORTC QLQH18. The investigators will ask each patient to answer to these questionnaires 6 months after treatment completion
Overall response rate based on the MRI evaluation in Child Pugh B7 patients | 6 months
  As the choice of the irradiation scheme will be influenced by the severity of the underlying cirrhosis with a Child Pugh score B7, the overall response rate in this specific kind of patients will be separately measured besides the overall response rate of the whole cohort.

OTHER OUTCOMES:
Immuno-histochemical detection of tumoral markers on biopsy (AFP/CK19/DCP) | at time of biopsy
  Differents markers will be checked on biopsy (AFP = alpha foetoprotein/ CK19 = cytokeratin 19/ DPC= Des Carboxy prothrombin).
Baseline biological detection of tumoral marker(s) : AFP +/- DCP | at baseline
  Biological detection of tumoral marker(s) will be done for every patient included in this trial (at least for AFP = alpha fetoprotein) at baseline then repeated every 2 months after treatment, up to 6 months. Measurement of DCP (Des-Carboxy-prothrombin will not be mandatory).
Biological detection of tumoral marker(s) (AFP +/- DCP) at 2 months after treatment | 2 months after treatment completion
  Biological detection of tumoral marker(s) will be done for every patient included in this trial (at least for AFP = alpha fetoprotein) at baseline then repeated every 2 months after treatment, up to 6 months. Measurement of DCP (Des-Carboxy-prothrombin will not be mandatory).
Biological detection of tumoral marker(s) (AFP +/- DCP) at 4 months after treatment | 4 months after treatment completion
  Biological detection of tumoral marker(s) will be done for every patient included in this trial (at least for AFP = alpha fetoprotein) at baseline then repeated every 2 months after treatment, up to 6 months. Measurement of DCP (Des-Carboxy-prothrombin will not be mandatory).
Biological detection of tumoral marker(s) (AFP +/- DCP) at 6 months after treatment | 6 months after treatment completion
  Biological detection of tumoral marker(s) will be done for every patient included in this trial (at least for AFP = alpha fetoprotein) at baseline then repeated every 2 months after treatment, up to 6 months. Measurement of DCP (Des-Carboxy-prothrombin will not be mandatory).
MRI description of tumors at the hepatobiliary phase at baseline | at baseline
  immunohistochemical markers and imaging features in hepatobiliary phase will be compared to see if any correlation can be detected
MRI description of tumors at the hepatobiliary phase at 2 months after treatment | 2 months after treatment completion
  immunohistochemical markers and imaging features in hepatobiliary phase will be compared to see if any correlation can be detected
MRI description of tumors at the hepatobiliary phase at 6 months after treatment | 6 months after treatment completion
  immunohistochemical markers and imaging features in hepatobiliary phase will be compared to see if any correlation can be detected

CONTACTS AND LOCATIONS:
Overall Officials: Xavier GEETS, Principal Investigator — Cliniques Universitaires Saint Luc/MIRO; Ivan BORBATH, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (5):
- Belgium (5):
  - Hôpital de JOLIMONT, Jolimont, Hainaut
  - Centre Hospitalier Universitaire/CHC Saint Joseph, Liège, Liège
  - Cliniques Universitaires Saint Luc, Brussels, Woluwé Saint Lambert
  - Institut Jules Bordet/Hôpital Erasme, Brussels
  - Clinique et Maternité Sainte Elisabeth/CHU Mont Godinne, Namur

IPD SHARING:
Plan to Share IPD: No
Every participant data will be anonymized for the trial purpose.